CLINICAL TRIAL: NCT01349153
Title: Facebook-based Physical Activity Intervention for Young Adult Cancer Survivors: the FITNET Randomized Pilot Study
Acronym: FITNET
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-2150
Record Dates: First submitted 2011-05-02; First posted 2011-05-06 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Physical Activity
Keywords: Physical Activity; Young Adults; Cancer Survivors
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Facebook-based Self-help Comparison (Active Comparator): Participants will receive a pedometer and twelve weekly messages with links to Internet resources that have educational materials related to exercise and cancer survivorship.
  Interventions: Behavioral: Facebook-based Self-help Comparison
- Facebook-based Messages/Website (Experimental): Participants will receive a pedometer, twelve weekly messages, and be encouraged to participate in sixteen Facebook group discussions and use a website for exercise goal-setting and tracking activity.
  Interventions: Behavioral: Facebook-based Messages/Website

INTERVENTIONS:
Behavioral: Facebook-based Messages/Website — Twelve weekly messages, a pedometer, sixteen group discussions, and access to an exercise website to promote increased physical activity.
  Arms: Facebook-based Messages/Website
Behavioral: Facebook-based Self-help Comparison — Twelve weekly messages and a pedometer.
  Arms: Facebook-based Self-help Comparison

SUMMARY:
The purpose of this study is to determine the feasibility and efficacy of a behavioral intervention, delivered through an existing social networking website (Facebook), on physical activity (moderate-intensity minutes per week) among young adult cancer survivors compared to a self-help education condition. For this research study, investigators will conduct a 12-week randomized trial. After a baseline survey, weekly messages, a pedometer, goal-setting tool, physical activity log and discussion prompts will be delivered to the intervention group. Comparison group participants will receive links to websites with self-help education materials. After 12 weeks, a follow-up survey will be given to both groups. Changes in physical activity, quality of life and psychosocial factors will be examined. The investigators hypothesize that those receiving the intervention will have improved physical activity behaviors at 12-week follow-up relative to those in the comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Young adult between ages 21-39 diagnosed with cancer (excluding non-melanoma skin cancer) at age 18 or older
* At least 1 year beyond date of diagnosis with no evidence of progressive disease or second primary cancers
* Completed cancer treatment
* English-speaking and writing
* No pre-existing medical condition(s) or contraindications that preclude adherence to an unsupervised exercise program, including cardiovascular disease, congestive heart failure, pulmonary conditions, renal disease, and severe orthopedic conditions
* Not adhering to the American Cancer Society's recommendation of at least 150 minutes of moderate-intensity exercise per week (<150 minutes/week)
* Have access to Internet service and an active Facebook account
* Willing to be randomized
* Have indicated consent by checking "yes" to the online consent form

Exclusion Criteria:

* Non-English speaking
* < 21 and > 39 years of age
* Diagnosed with cancer less than one year previously or still in treatment
* Pre-existing medical condition(s) that preclude adherence to an unsupervised exercise program, including cardiovascular disease, congestive heart failure, pulmonary conditions, renal disease, and severe orthopedic conditions

Ages: 21 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Primary study outcome measures at the participant level will be minutes of moderate-intensity physical activity per week and exercise in MET-hrs/week. | Participants will be assessed at baseline (before 12-week study period) and after 12 weeks.

SECONDARY OUTCOMES:
Quality of life | Participants will be assessed at baseline (before 12-week study period) and after 12 weeks.
Psychosocial factors | Participants will be assessed at baseline (before 12-week study period) and after 12 weeks.
  Examine potential mediators of the effect of the intervention, including changes in self-efficacy, social support and self-monitoring behaviors
Utilization of program components/activities | Participants will be assessed at baseline (before 12-week study period) and after 12 weeks.
Perceptions of program components/activities | Participants will be assessed at baseline (before 12-week study period) and after 12 weeks.
Communication factors | Participants will be assessed at baseline (before 12-week study period) and after 12 weeks.
  Examine potential mediators of the effect of the intervention, including message trust, relevance and recall

CONTACTS AND LOCATIONS:
Overall Officials: Marci K. Campbell, PhD, MPH, Study Chair — University of North Carolina, Chapel Hill; Carmina G. Valle, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Lineberger Comprehensive Cancer Center at UNC-CH, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Valle CG, Tate DF. Engagement of young adult cancer survivors within a Facebook-based physical activity intervention. Transl Behav Med. 2017 Dec;7(4):667-679. doi: 10.1007/s13142-017-0483-3. PMID 28374211
- [Derived] Valle CG, Tate DF, Mayer DK, Allicock M, Cai J. A randomized trial of a Facebook-based physical activity intervention for young adult cancer survivors. J Cancer Surviv. 2013 Sep;7(3):355-68. doi: 10.1007/s11764-013-0279-5. Epub 2013 Mar 27. PMID 23532799